CLINICAL TRIAL: NCT03965182
Title: A Head-to-head Comparison Study of Polyethylene Glycol, Polyethylene Glycol Plus Sodium Picosulfate, and Sodium Picosulfate
Brief Title: Compare Polyethylene Glycol and Sodium Picosulfate Alone or Combined
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: A10801001
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-04

CONDITIONS: Bowel Preparation
Keywords: colon preparation, ,; polyethylene glycol; sodium picosulfate/magnesium citrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PEG group (Active Comparator): Patients in the PEG group were instructed to take the first sachet of PEG at 19:00 hours the day before colonoscopy and the second one at 06:00 hours on the morning of the day of colonoscopy.
  Interventions: Drug: PEG
- PEG plus SPMC group (Active Comparator): Patients in the PEG plus SPMC group will be instructed to take the SPMC sachet at 19:00 hours the day before colonoscopy and the PEG sachet at 6:00 hours on the morning of the day of colonoscopy.
  Interventions: Drug: PEG plus SPMC
- SPMC group (Active Comparator): Patients in the SPMC group were instructed to take the first sachet of SPMC at 19:00 hours the day before colonoscopy and the second one at 06:00 hours on the morning of the day of colonoscopy.
  Interventions: Drug: SPMC

INTERVENTIONS:
Drug: PEG — 2 sachets of PEG will be used as the bowel prep regimen.
  Arms: PEG group
Drug: PEG plus SPMC — one sachet of PEG and one sachet will be administered as the bowel prep regimen
  Arms: PEG plus SPMC group
Drug: SPMC — 2 sachets will be administered as the bowel prep regimen.
  Arms: SPMC group

SUMMARY:
Sodium picosulfate/magnesium citrate (SPMC) is generally better tolerated than PEG, its cleansing effect remains uncertain. While most studies showed SPMC was non-inferior to PEG, some studies reported that SPMC was less effective than PEG. To improve the bowel cleansing effect of SPMC, splitting the dose by using one sachet the evening before colonoscopy and the other sachet 4 to 5 hours before colonoscopy in the morning, has been proposed.Adding bisacodyl to the regimen also has been shown to be helpful. Some side effects, such as hyponatremia, dehydration and sleep disturbance, were reported to be more commonly associated with SPMC than with PEG.

To enhance the efficacy and reduce the side effects, two studies have evaluated the combination of SPMC and PEG, with conflicting results.The effect of combining PEG and SPMC should be best appreciated with head-to-head comparison with PEG and SPMC alone at the same time.

Therefore we designed this head-to-head comparison study for 2 L PEG, 1L PEG plus one sachet of SPMC and 2 sachet of SPMC, all with split-dose and the addition of 10 ml bisacodyl. Our hypothesis is the bowel cleansing effect of the combination regimen was not inferior to PEG alone. The tolerability, acceptability and side effects of the 3 regimen will also be evaluated.

Patients will be randomly assigned to either PEG, PEG plus SPMC or SPMC group, in a 1:1:1 ratio using a computer-generated sequence. The treatment allocation will be concealed and revealed by non-research medical personnel at the screening visit.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will include those anticipated to undergo colonoscopy, aged 20 to 80 at the time of enrollment.

Exclusion Criteria:

* previous colon resection, gastrointestinal obstruction, ileus, intestinal perforation, toxic megacolon, active stage of inflammatory bowel disease, congestive heart failure (New York Heart Association Class III or IV),acute cardiovascular disease, uncontrolled arterial hypertension (systolic pressure >170 mmHg, diastolic pressure>100 mmHg), severe liver cirrhosis (Child-Pugh score C) or renal failure (creatinine clearance<30 mL/minute) or any allergy to, PEG, or sodium picosulfate solution, phenylketonuria, and glucose-6-phosphate dehydrogenase deficiency.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Aronchick scale | through study completion, average 30 minutes
  a validated assessment that describes the visual appearance of the colon on a four-point scale.
Boston Bowel Preparation Scale | through study completion, average 30 minutes
  BBPS is based on the summation of the preparation scores from three segments of the colon (cecum and ascending, transverse colon and left colon). A segment score of 0 describes an"unprepared colon segment with mucosa not well seen due to solid stool that cannot be cleared"; segment score 1: "portion of mucosa of the colon segment seen, but other areas of the colon are not well seen due to staining, residual stool and⁄or opaque liquid"; segment score 2: "minor amount of residual staining, small fragments of stool and⁄or opaque liquid, but mucosa of colon segment seen well"; segment score 3: "entire mucosa of the colon segment seen well with no residual staining, small fragments of stool and⁄or opaque liquid".

SECONDARY OUTCOMES:
Adenoma detection rate | when pathology of polyps become available, average in one week.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsi Hsieh, MD, Principal Investigator — Buddhist Dalin Tzu Chi Hospital

REFERENCES:
- [Background] Froehlich F, Wietlisbach V, Gonvers JJ, Burnand B, Vader JP. Impact of colonic cleansing on quality and diagnostic yield of colonoscopy: the European Panel of Appropriateness of Gastrointestinal Endoscopy European multicenter study. Gastrointest Endosc. 2005 Mar;61(3):378-84. doi: 10.1016/s0016-5107(04)02776-2. PMID 15758907
- [Background] Harewood GC, Sharma VK, de Garmo P. Impact of colonoscopy preparation quality on detection of suspected colonic neoplasia. Gastrointest Endosc. 2003 Jul;58(1):76-9. doi: 10.1067/mge.2003.294. PMID 12838225
- [Background] Rex DK, Imperiale TF, Latinovich DR, Bratcher LL. Impact of bowel preparation on efficiency and cost of colonoscopy. Am J Gastroenterol. 2002 Jul;97(7):1696-700. doi: 10.1111/j.1572-0241.2002.05827.x. PMID 12135020
- [Background] Enestvedt BK, Tofani C, Laine LA, Tierney A, Fennerty MB. 4-Liter split-dose polyethylene glycol is superior to other bowel preparations, based on systematic review and meta-analysis. Clin Gastroenterol Hepatol. 2012 Nov;10(11):1225-31. doi: 10.1016/j.cgh.2012.08.029. Epub 2012 Aug 30. PMID 22940741
- [Background] Marshall JB, Pineda JJ, Barthel JS, King PD. Prospective, randomized trial comparing sodium phosphate solution with polyethylene glycol-electrolyte lavage for colonoscopy preparation. Gastrointest Endosc. 1993 Sep-Oct;39(5):631-4. doi: 10.1016/s0016-5107(93)70213-8. PMID 8224683
- [Background] Valiante F, Bellumat A, De Bona M, De Boni M. Bisacodyl plus split 2-L polyethylene glycol-citrate-simethicone improves quality of bowel preparation before screening colonoscopy. World J Gastroenterol. 2013 Sep 7;19(33):5493-9. doi: 10.3748/wjg.v19.i33.5493. PMID 24023492
- [Background] de Leone A, Tamayo D, Fiori G, Ravizza D, Trovato C, De Roberto G, Fazzini L, Dal Fante M, Crosta C. Same-day 2-L PEG-citrate-simethicone plus bisacodyl vs split 4-L PEG: Bowel cleansing for late-morning colonoscopy. World J Gastrointest Endosc. 2013 Sep 16;5(9):433-9. doi: 10.4253/wjge.v5.i9.433. PMID 24044042
- [Background] Clark RE, Godfrey JD, Choudhary A, Ashraf I, Matteson ML, Bechtold ML. Low-volume polyethylene glycol and bisacodyl for bowel preparation prior to colonoscopy: a meta-analysis. Ann Gastroenterol. 2013;26(4):319-324. PMID 24714413
- [Background] Katz PO, Rex DK, Epstein M, Grandhi NK, Vanner S, Hookey LC, Alderfer V, Joseph RE. A dual-action, low-volume bowel cleanser administered the day before colonoscopy: results from the SEE CLEAR II study. Am J Gastroenterol. 2013 Mar;108(3):401-9. doi: 10.1038/ajg.2012.441. Epub 2013 Jan 15. PMID 23318484
- [Background] Rex DK, Katz PO, Bertiger G, Vanner S, Hookey LC, Alderfer V, Joseph RE. Split-dose administration of a dual-action, low-volume bowel cleanser for colonoscopy: the SEE CLEAR I study. Gastrointest Endosc. 2013 Jul;78(1):132-41. doi: 10.1016/j.gie.2013.02.024. Epub 2013 Apr 6. PMID 23566639
- [Background] Kim HG, Huh KC, Koo HS, Kim SE, Kim JO, Kim TI, Kim HS, Myung SJ, Park DI, Shin JE, Yang DH, Lee SH, Lee JS, Lee CK, Chang DK, Joo YE, Cha JM, Hong SP, Kim HJ. Sodium Picosulfate with Magnesium Citrate (SPMC) Plus Laxative Is a Good Alternative to Conventional Large Volume Polyethylene Glycol in Bowel Preparation: A Multicenter Randomized Single-Blinded Trial. Gut Liver. 2015 Jul;9(4):494-501. doi: 10.5009/gnl14010. PMID 25287163
- [Background] Gweon TG, Kim SW, Noh YS, Hwang S, Kim NY, Lee Y, Lee SW, Lee SW, Lee JY, Lim CH, Hun Kim H, Kim JS, Kyung Cho Y, Myung Park J, Seok Lee I, Myung-Gyu Choi. Prospective, randomized comparison of same-day dose of 2 different bowel cleanser for afternoon colonoscopy: picosulfate, magnesium oxide, and citric acid versus polyethylene glycol. Medicine (Baltimore). 2015 Apr;94(13):e628. doi: 10.1097/MD.0000000000000628. PMID 25837751
- [Background] Manes G, Amato A, Arena M, Pallotta S, Radaelli F, Masci E. Efficacy and acceptability of sodium picosulphate/magnesium citrate vs low-volume polyethylene glycol plus ascorbic acid for colon cleansing: a randomized controlled trial. Colorectal Dis. 2013 Sep;15(9):1145-53. doi: 10.1111/codi.12246. PMID 23581277
- [Background] Dakkak M, Aziz K, Bennett JR. Short report: comparison of two orally administered bowel preparations for colonoscopy--polyethylene glycol and sodium picosulphate. Aliment Pharmacol Ther. 1992 Aug;6(4):513-9. doi: 10.1111/j.1365-2036.1992.tb00566.x. PMID 1420744
- [Background] Jin Z, Lu Y, Zhou Y, Gong B. Systematic review and meta-analysis: sodium picosulfate/magnesium citrate vs. polyethylene glycol for colonoscopy preparation. Eur J Clin Pharmacol. 2016 May;72(5):523-32. doi: 10.1007/s00228-016-2013-5. Epub 2016 Jan 28. PMID 26818765
- [Background] Klare P, Poloschek A, Walter B, Rondak IC, Attal S, Weber A, von Delius S, Bajbouj M, Schmid RM, Huber W. Single-day sodium picosulfate and magnesium citrate versus split-dose polyethylene glycol for bowel cleansing prior to colonoscopy: A prospective randomized endoscopist-blinded trial. J Gastroenterol Hepatol. 2015 Nov;30(11):1627-34. doi: 10.1111/jgh.13010. PMID 25968966
- [Background] Flemming JA, Vanner SJ, Hookey LC. Split-dose picosulfate, magnesium oxide, and citric acid solution markedly enhances colon cleansing before colonoscopy: a randomized, controlled trial. Gastrointest Endosc. 2012 Mar;75(3):537-44. doi: 10.1016/j.gie.2011.09.018. Epub 2011 Dec 21. PMID 22192423
- [Background] Hookey LC, Vanner SJ. Pico-salax plus two-day bisacodyl is superior to pico-salax alone or oral sodium phosphate for colon cleansing before colonoscopy. Am J Gastroenterol. 2009 Mar;104(3):703-9. doi: 10.1038/ajg.2008.167. Epub 2009 Feb 17. PMID 19223885
- [Background] Labuschagne GS, Morris RW. The effect of oral intake during the immediate pre-colonoscopy time period on volume depletion in patients who receive sodium picosulfate. Anaesth Intensive Care. 2017 Jul;45(4):485-489. doi: 10.1177/0310057X1704500412. PMID 28673219
- [Background] Sharara AI, El Reda ZD, Harb AH, Abou Fadel CG, Sarkis FS, Chalhoub JM, Abou Mrad R. The burden of bowel preparations in patients undergoing elective colonoscopy. United European Gastroenterol J. 2016 Apr;4(2):314-8. doi: 10.1177/2050640615594550. Epub 2015 Jul 3. PMID 27087962
- [Background] Weir MA, Fleet JL, Vinden C, Shariff SZ, Liu K, Song H, Jain AK, Gandhi S, Clark WF, Garg AX. Hyponatremia and sodium picosulfate bowel preparations in older adults. Am J Gastroenterol. 2014 May;109(5):686-94. doi: 10.1038/ajg.2014.20. Epub 2014 Mar 4. PMID 24589671
- [Background] Kim MJ, Hong CW, Kim BC, Park SC, Han KS, Joo J, Oh JH, Sohn DK. Phase II Randomized Controlled Trial of Combined Oral laxatives Medication for BOwel PREParation (COMBO-PREP study). Medicine (Baltimore). 2016 Feb;95(7):e2824. doi: 10.1097/MD.0000000000002824. PMID 26886637
- [Background] Song KH, Suh WS, Jeong JS, Kim DS, Kim SW, Kwak DM, Hwang JS, Kim HJ, Park MW, Shim MC, Koo JI, Kim JH, Shon DH. Effectiveness of Sodium Picosulfate/Magnesium Citrate (PICO) for Colonoscopy Preparation. Ann Coloproctol. 2014 Oct;30(5):222-7. doi: 10.3393/ac.2014.30.5.222. Epub 2014 Oct 28. PMID 25360429